CLINICAL TRIAL: NCT05216900
Title: Breast Reconstruction and Neoadjuvant Therapy, a Changing Algorithm
Brief Title: Breast Reconstruction and Neoadjuvant Radiotherapy
Acronym: BRENAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Alexander Monro Hospital, Bilthoven (Unknown); Amsterdam UMC (Other); Cancer Center Amsterdam grant for innovative research (Unknown)
Responsible Party: Principal Investigator, Wiesje Maarse, Principal investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80252
Record Dates: First submitted 2021-12-28; First posted 2022-02-01 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Neoadjuvant radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a prospective multicenter single arm interventional pilot study. The primary endpoint is post-surgical complications at three months after the latest patient has received the final reconstructive surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant radiotherapy group (Experimental): Twenty breast cancer patients will be included after they have given informed consent. Patients are eligible if they have an indication for mastectomy and RT, and a wish for an immediate reconstruction, either implant-based or autologous, in UMCU, Alexander Monro hospital, St Antonius Hospital, ZiekenhuisGroep Twente, Haagladen Medical Center and Amsterdam UMC.
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — The study examines the delivery NART.
  In case of neoadjuvant chemotherapy, RT will start 6-8 weeks after the last course of chemotherapy. A dose of 15 x 2.67 Gy 5 fractions per week, or a biologically equivalent dose will be applied.
  A mastectomy and a direct breast reconstruction will be performed, approximately 2-6 weeks after latest radiotherapy treatment. Breast reconstruction can be separated in the types of reconstruction, either reconstruction with a silicone implant or with only autologous tissue, of which the most common flap used is the Deep Inferior Epigastric Perforator (DIEP) flap.

SUMMARY:
The purpose the BRENAR pilot study is to assess acute post-surgical complications following mastectomy and immediate breast reconstruction after neoadjuvant radiotherapy (NART). The investigators hypothesize that NART will avoid the negative effects of postmastectomy radiotherapy (PMRT) on the capsule of an implant, or on the skin and underlying tissue of an autologous flap, and would therefore lead to better cosmetic results, better quality of life and less complications compared to PMRT. If this hypothesis is confirmed, NART would allow more patients to undergo an immediate reconstruction resulting in superior cosmetic results and quality of life. Furthermore, the use of RT in a neoadjuvant setting could potentially result in a shorter overall loco-regional treatment time from diagnosis to receiving the last locoregional treatment. However, this pilot study will mainly assess whether or not the post-surgical complications of breast reconstruction with NART are acceptable. Further study to investigate long term quality of life and oncologic follow-up results will be conducted after this pilot study, if complication rates are acceptable.

DETAILED DESCRIPTION:
Rationale: Treatment of patients with breast cancer requires a multimodality approach with often systemic therapy, radiotherapy (RT) and surgery. Postmastectomy radiotherapy (PMRT) reduces locoregional recurrences and improves survival, especially in patients with involved axillary nodes. However, PMRT is known to substantially increase the complication rate when combined with a breast reconstruction. Breast reconstructions can be performed within the same surgery as the mastectomy (i.e. immediate) or in a later stage where patients remain without a breast contour for several months to years before the reconstruction is completed (i.e. delayed).

In the Netherlands, most patients are being withheld an immediate breast reconstruction if there is the slightest risk of PMRT, because PMRT in combination with immediate breast reconstruction is associated with a severe increase in postoperative complications, especially in case of an implant-based reconstruction: complication rates up to 40% have been reported, in comparison to less than 10% without PMRT. Short-term complications include infection and loss of implant, while long-term complications include pain, capsular contracture and fibrosis. Such complications have been shown to negatively affect quality of life, perceived body image and sexual well-being. Furthermore, PMRT after an immediate reconstruction is associated with impaired cosmetic results and lower patient satisfaction, even when no complications have occurred.

If patients aim for an autologous reconstruction (i.e. use of own tissue), usually PMRT is performed first, followed by a delayed autologous reconstruction to avoid radiotherapy on the flap, thereby subjecting patients to a second major surgical procedure and a long period of living without a breast contour.

The unsatisfying cosmetic results and high complication rate have led to controversy and a wide practice variation in reconstruction approaches that are being offered to this specific group of patients. Since immediate breast reconstructions have proven to yield better cosmetic outcomes, psychosocial results and reduced overall costs, solutions that would allow for an immediate breast reconstruction in combination with radiation therapy (RT), without an increase in complications, are highly needed. Previous studies in breast cancer patients indicated that neoadjuvant RT (NART) is a safe approach from an oncological perspective, and does not increase the overall post-operative complication rate. However, limited data are available on NART in combination with an immediate breast reconstruction, and no data are available on patient-reported cosmetic outcomes.

Objective: The purpose of the pilot study is to assess acute post-surgical complications following mastectomy and immediate breast reconstruction after NART. The investigators hypothesize that NART will avoid the negative effects of PMRT on the capsule of an implant, or on the skin and underlying tissue of an autologous flap, and would therefore lead to better cosmetic results, better quality of life and less complications compared to PMRT. If this hypothesis is confirmed, NART would allow more patients to undergo an immediate reconstruction resulting in superior cosmetic results and quality of life. Furthermore, the use of RT in a neoadjuvant setting could potentially result in a shorter overall loco-regional treatment time from diagnosis to receiving the last locoregional treatment. However, this pilot study will mainly assess whether or not the post-surgical complications of breast reconstruction with NART are acceptable. Further study to investigate long term quality of life and oncologic follow-up results will be conducted after this pilot study, if complication rates are acceptable.

Study design: The study will be conducted as a prospective multicenter single arm interventional pilot study. The primary endpoint is post-surgical complications at three months after the latest patient has received the final reconstructive surgery.

Study population: Twenty breast cancer patients will be included after they have given informed consent. Patients are eligible if they have an indication for mastectomy and RT, and a wish for an immediate reconstruction, either implant-based or autologous, in MUMC, UMCU, Alexander Monro hospital and Amsterdam UMC.

Intervention (if applicable): The intervention consists of NART followed by mastectomy with immediate reconstruction, where the standard treatment is mastectomy and PMRT, with an immediate or delayed reconstruction.

Main study parameters/endpoints:

Primary endpoint: Acute post-surgical complications at 3 months following mastectomy and immediate breast reconstruction after NART in the treatment of breast cancer.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Burden:

Currently, in certain hospitals, the indication for RT is based upon the pathological nodal status of the sentinel or previously involved nodes, removed during mastectomy. Since patients in this study will receive NART, the indication for RT is not always clear prior to surgery. In those cases, an axillary staging procedure has to be performed prior to the breast surgery, to determine whether there is an indication for RT at all. This requires two separate surgical procedures, which is nowadays already common practice in several hospitals, to determine whether an immediate breast reconstruction is possible. Currently, for cT1-3N0 patients, it is known that about 25% has a positive axillary node after neoadjuvant chemotherapy and thus still requires PMRT; for patients with cT1-3N+ breast cancer, about 55-70% still have positive nodes after neoadjuvant chemotherapy requiring PMRT. Consequently, some patients that have given their informed consent for NART but will be excluded from this study if the sentinel node appears to be free of tumor cells.

Another additional burden can be an additional biopsy of the tumor after neoadjuvant chemotherapy, to determine whether residual disease is present. If residual disease is present, there is also an indication for adjuvant systemic treatment in triple negative patients or her2- positive patients. Since a biopsy is not sufficiently accurate to determine pCR status, patients are excluded from the study if the biopsy does not contain tumors cells, since NART can influence the final pathological tumor status.

Finally, from a patient's perspective, additional time is required for filling in questionnaires with regard to cosmetic results and quality of life (approximately 15-30 minutes).

Risk Data from current pilot studies indicates that NART is at least as effective as PMRT with regard to oncologic safety. A risk that is associated with participation is the possibility of decreased vascularization of the skin (nipple) flap of the breast after a sparing mastectomy leading to early complications, especially in the implant group. However, it is anticipated that this risk of necrosis and loss of tissue expander/implant is low, since previous pilot studies showed that overall short and long-term complications were similar between PMRT and NART.

Benefit and group relatedness:

NART will allow patients to always receive an immediate breast reconstruction (both implant-based and autologous), even is RT is indicated. It is hypothesized that this will result in a better QoL and cosmetic outcome. Finally total treatment time will be shorter with NART.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:
* Females at least 18 years of age.
* WHO performance scale ≤2
* Adequate communication and understanding skills of the Dutch language
* Able to understand and sign Dutch written informed consent
* Indication for mastectomy and a known indication for (adjuvant) radiotherapy of at least the chestwall. To obtain information on the indication for RT, before the mastectomy is performed, it may be necessary to perform a separate SNP and/or targeted axillary dissection prior to inclusion, i.e.

  * Stage III (cT3N1, cT0-2N2-3) or cN1 with more than 3 suspicious nodes at initial diagnosis
  * A positive SN/TAD* pre- breast surgery in case of:
* cT1-2N0 and less than 3 RF** at initial diagnosis and cCR on imaging***
* cT3N0 and no risk factor at initial diagnosis

  * If the indication for radiotherapy is not yet clear, and is only indicated when there is a pathological lymph node present, a sentinel node procedure or targeted axillary dissection (TAD) will be performed first to check for the lymph node status. A sentinel node procedure (SNP) will be performed under general anesthesia in order to explore regional lymph nodes. For cT1-3N0 patients, it is known that about 25% has a positive axillary node after neoadjuvant chemotherapy (50);for patients with cT1-3N+ breast cancer, about 55-70% still have positive nodes after neoadjuvant chemotherapy, which is dependent of receptor status 29,30,31,32,33. Consequently, we may have to ask for informed consent 2-4 times more patients than we would need for this pilot study.

    * risk factors are: angio invasion, Grade III, Age ≤ 40 yrs, triple negative *** In patients with cT1-2N0 with at least 3 RF a tumour biopsy can be considered prior to surgery in case of neoadjuvant chemotherapy, since in case of no pCR the indication for RT is already set, and an SN or TAD prior to breast surgery is not required.

Exclusion Criteria:

* study:
* Legal incapacity
* Not able to understand and sign Dutch written informed consent
* Previous history of breast cancer or another malignancy for which radiotherapy of the breast or axilla
* Collagen synthesis disease
* MRI absolute contraindications as defined by the Radiology Department
* Age < 18 year
* Pregnant or lactating.
* Smoking
* BMI > 35 kg/m2
* cT4 tumour (and skin sparing mastectomy not possible)
* If NAC in cT1-2N0 and 3 RF: in triple negative or Her2 positive (with concern for under treatment of adjuvant therapy) and no tumor cells in preoperative biopsy*

  * NB: If neoadjuvant chemotherapy is given, and if the indication for adjuvant systemic treatment is dependent on the presence or absence of a pathological complete response pCR (such as in patients with a triple negative or Her2 positive tumour), centres can choose A) to exclude these patients, or B) only to include these patients when a non-pCR is proven via a biopsy prior to the start of the RT. Earlier studies in partial breast RT showed that pCR rate of NART only, followed by surgery < 6-8 weeks is very low in the general breast cancer population (17 of the 110), whilst it seems to be higher in patients with triple negative (6/8) and Her2 positive (1/1) (personal communication Sophie Bosma, trial on Preoperative Accelerated Partial Breast Irradiation, PAPBI trial 34.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Acute post-surgical complication rate at 3 months following mastectomy and immediate breast reconstruction after NART in the treatment of breast cancer. | 3 months following mastectomy and immediate breast reconstruction (latest intervention, being either autologous recosntruction or silicone implant)
  Surgical complications are defined as any complication requiring surgical intervention necessary (excluding percutaneous drainage and antibiotic treatment for inflammation in cases without need for open drainage) within a period up to three months after the final reconstruction, defined and scored using the Clavien-Dindo Classification of Surgical Complications (C-DC)37: - Infection - Hematoma - Loss of implant/expander/flap - (Fat)Necrosis

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Within 3 months after both breast reconstruction and radiotherapy
  Other adverse events following NART or surgery other than described in the primary outcome measure.
Patient-reported Satisfaction with Breasts, Physical, emotional and sexual well-being (as measured using BREAST-Q) | At baseline and 3 months after definitive treatment (definitive breast reconstruction).
  The BREAST-Q is a multiscale, multimodule, patient-reported outcome instrument measuring important aspects of health-related quality of life and patient satisfaction in women who undergo breast surgery.The BREAST-Q has multiple domains, and each domain score is obtained by transforming the raw scale item responses with the Q-Score software program. Each domain results in an independent score from 0 to 100 (higher scores indicate greater satisfaction or quality of life).
The Aesthetic Items Scale; Physician-reported cosmetic results of the reconstructed breast | 3 months after definitive breast reconstruction surgery
  The clinical investigators will assess the physician-reported aesthetic outcome from photographs using the Aesthetic Items Scale,12 which is a standardised method*. Five standardised photographs will be taken before and at 3 months after placement of the breast implant. The photos will be evaluated independently by five plastic surgeons. The surgeons will rate the aesthetic outcome on five items with a five-point Likert scale12. The breasts are evaluated with respect to volume, shape, symmetry, scars, and nipple areola complex. For each of these items a 5-point Likert scale is used for scoring. This scale ranges from "very dissatisfied," "dissatisfied," "neutral," "satisfied," to "very satisfied."
  The summed score of the 5 items as the Total Aesthetic Score (TAS) with high scores meaning better outcome.
  * Dikmans et al. The Aesthetic Items Scale: A Tool for the Evaluation of Aesthetic Outcome after Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Mar 1;5(3)
Timely initiation of (possible) adjuvant therapy | In three months after mastectomy
Pathological complete response (pCR) assessed in mastectomy specimen | Within 2 weeks after mastectomy
  A pCR was defined as absence of invasive and in situ carcinoma in the breast, irrespective of nodal status (ypT0). Response of the breast was assessed according to EUSOMA.
  1. Complete pathological response, either (i) no residual carcinoma or (ii) no residual invasive carcinoma but DCIS present.
  2. Partial response to therapy, either (i) minimal residual disease/near total effect (e.g. only a few loose tumour cells or tumour cells located in small groups) or (ii) evidence of response to therapy but with 10-50% of tumour remaining or (iii) >50% of tumour cellularity remains evident, when compared to the previous core biopsy sample, although some features of response to therapy are present (e.g. fibrosis).
  3. No response: no evidence of response to therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Maarse Wiesje, Bilthoven, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No